CLINICAL TRIAL: NCT06593730
Title: Double-blind, Placebo-controlled, Randomised, Parallel-group Study in Healthy Volunteers to Evaluate the Safety, Tolerability, Pharmacodynamic Effects and Pharmacokinetics of Twice Daily Intra-anal Application of NRL001-cream for 14 Days.
Brief Title: Safety and Tolerability of the Twice Daily Intra-anal Application of NRL001 Cream for 14 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NRL001-01/2007(RD)
Record Dates: First submitted 2015-06-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Faecal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- NRL001 cream 0.5%w/w (Experimental): 0.5%w/w NRL001 (1R,2S-methoxamine) 1 mL, twice daily administration (morning and afternoon) for 14 days (study Days D1 to D14).
  Interventions: Drug: NRL001 cream 0.5%w/w
- NRL001 cream 0.75% w/w (Experimental): 0.75%w/w NRL001 (1R,2S-methoxamine) 1 mL, twice daily administration (morning and afternoon) for 14 days (study Days D1 to D14).
  Interventions: Drug: NRL001 cream 0.75%w/w
- NRL001 cream 1.0% w/w (Experimental): 1.0%w/w NRL001 (1R,2S-methoxamine) 1 mL, twice daily administration (morning and afternoon) for 14 days (study Days D1 to D14).
  Interventions: Drug: NRL001 cream 1.0%w/w
- NRL001 cream 1.5% w/w (Experimental): 1.5%w/w NRL001 (1R,2S-methoxamine) 1 mL, twice daily administration (morning and afternoon) for 14 days (study Days D1 to D14).
  Interventions: Drug: NRL001 cream 1.5%w/w
- NRL001 cream 2.0% w/w (Experimental): 2.0%w/w NRL001 (1R,2S-methoxamine) 1 mL, twice daily administration (morning and afternoon) for 14 days (study Days D1 to D14).
  Interventions: Drug: NRL001 cream 2.0%w/w
- NRL001 cream 2.5% w/w (Experimental): 2.5%w/w NRL001 (1R,2S-methoxamine) 1 mL, twice daily administration (morning and afternoon) for 14 days (study Days D1 to D14).
  Interventions: Drug: NRL001 cream 2.5%w/w

INTERVENTIONS:
Drug: NRL001 cream 0.5%w/w
  Other Names: NRL001 (1R,2S-methoxamine) cream 0.5%w/w
  Arms: NRL001 cream 0.5%w/w
Drug: NRL001 cream 0.75%w/w
  Other Names: NRL001 (1R,2S-methoxamine) cream 0.75%w/w
  Arms: NRL001 cream 0.75% w/w
Drug: NRL001 cream 1.0%w/w
  Other Names: NRL001 (1R,2S-methoxamine) cream 1.0%w/w
  Arms: NRL001 cream 1.0% w/w
Drug: NRL001 cream 1.5%w/w
  Other Names: NRL001 (1R,2S-methoxamine) cream 1.5%w/w
  Arms: NRL001 cream 1.5% w/w
Drug: NRL001 cream 2.0%w/w
  Other Names: NRL001 (1R,2S-methoxamine) cream 2.0%w/w
  Arms: NRL001 cream 2.0% w/w
Drug: NRL001 cream 2.5%w/w
  Other Names: NRL001 (1R,2S-methoxamine) cream 2.5%w/w
  Arms: NRL001 cream 2.5% w/w

SUMMARY:
The study is being conducted to evaluate the safety and tolerability after single and repeated twice daily intra-anal applications of 1mL NRL001 cream in stepwise increasing concentrations.

DETAILED DESCRIPTION:
Single-centre, randomised, placebo-controlled, double-blind, repeated dose study in healthy male and female volunteers, comprising up to six sequential dose groups receiving 1 mL doses of an investigational cream formulation containing 0.50, 0.75, 1.00, 1.50, 2.00 and 2.50% w/w NRL001. Doses were to be investigated in stepwise increasing fashion. Progression to a higher dose-step required completion of the previous dose-step without safety limiting findings. Each dose-step was to be investigated in 12 subjects; in each dose-group, subjects assigned to active treatment were to be studied in parallel with subjects assigned to placebo in double-blind fashion with random (9:3) treatment assignment. Each subject was to be studied for one study period with double-blind investigational treatment (1 mL of an investigational cream formulation containing NRL001 or matched placebo) twice daily from the morning of D01 to the afternoon of D14; this phase was to be preceded by a single-blind placebo control day (D-1) with administration of placebo in the morning and afternoon.

ELIGIBILITY:
Inclusion Criteria:

* Males or females (only females of non-child-bearing potential or of child-bearing potential while taking medically appropriate contraception)
* Caucasian
* 35 to 60 years of age (included)
* BMI: between 22 and 26 kg.m-2
* BW: between 50 and 100 kg
* Willing and able to provide written informed consent

Exclusion Criteria:

General - all subjects

* Previous participation in the trial
* Participation in any other trial during the last 90 days
* Donation of blood or plasma within the last 90 days before recruitment
* History of any clinically relevant allergy
* Presence of acute or chronic infection
* Presence or history of any relevant medical condition or disease (as evaluated on the basis of medical history, physical examination, recumbent and standing blood pressure, treadmill ergometry, clinical laboratory tests [haematology, clinical chemistry, urinalysis, serology])
* Presence or history of migraine, frequent headaches, Raynaud phenomenon, urinary urge, signs and symptoms of prostatism
* Presence or history of regular/habitual diarrhoea or constipation; previous anal surgery or trauma, anal fissures, rectal disorders
* Resting systolic blood pressure > 145 or < 90 mmHg, diastolic blood pressure > 95 or < 50 mmHg
* Positive treadmill ergometry test
* Resting pulse (PR) or electrocardiographic heart rate (HR) < 55 bpm
* ECG: AV-block (AV-block grade I included), QT > 480 msec, QTc > 450 msec, sick-sinus syndrome
* Positive hepatitis (HBs-Ag or HBc-Ab, HCV-Ab) or HIV serology test
* History of alcohol or (social) drug abuse
* Positive alcohol or urine drug test
* Daily consumption of > 30 g alcohol
* Smoking more than 15 cigarettes/day or equivalent of other tobacco products
* Use of prohibited medication
* Suspicion or evidence that the subject is not reliable
* Suspicion or evidence that the subject is not able to make a free consent or to understand the information detailed in the Subject Information sheet.

All females

* Positive pregnancy test
* Lactating
* Premenopausal women : not using contraception which is judged adequate and sufficient in the opinion of the clinical investigator

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2007-08; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Recumbent and standing blood pressure and pulse rate | 17 days
  BP and pulse taken lying and standing at screening, on control day and profiling days
Ambulatory 24 hour BP monitoring | 17 days
  Ambulatory 24 hour BP monitoring on control day and profiling days
12-lead digital resting ECG | 17 days
  12-lead digital resting ECG at screening, on control day and profiling days
3-lead ambulatory 24 hour ECG monitoring | 17 days
  24 hour HOLTER monitoring at screening, on control day and profiling days

SECONDARY OUTCOMES:
Plasma concentrations of NRL001 | 17 days
  Single and repeat dose pharmacokinetics of NRL001 in plasma
Well being | 17 days
  Any untoward change in health and/or wellbeing
Adverse events | 17 days
  Any unwanted sign or symptom